CLINICAL TRIAL: NCT02379520
Title: HPV-16/18 E6/E7-Specific T Lymphocytes in Patients With Relapsed HPV-Associated Cancers
Brief Title: HPV-16/18 E6/E7-Specific T Lymphocytes, Relapsed HPV-Associated Cancers, HESTIA
Acronym: HESTIA
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Carlos Ramos, Assistant Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-36021 HESTIA
Record Dates: First submitted 2015-02-25; First posted 2015-03-05 (Estimated); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Human Papillomavirus-Related Carcinoma; Human Papillomavirus Positive Oropharyngeal Carcinoma; Human Papillomavirus Positive Cervical Carcinoma; Human Papillomavirus Positive Anal Carcinoma; Human Papillomavirus Positive Vulvar Carcinoma; Human Papillomavirus Positive Penile Carcinoma
Keywords: recurrent cancer; refractory cancer; virus specific T-cells; gene therapy; HPV
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): HPV Specific T Cells
  Interventions: Genetic: HPV Specific T Cells
- Group B (Experimental): HPV Specific T Cells plus lymphodepletion (Cytoxan and Fludarabine) and nivolumab
  Interventions: Genetic: HPV Specific T Cells; Drug: Cytoxan; Drug: Fludarabine; Biological: Nivolumab

INTERVENTIONS:
Genetic: HPV Specific T Cells — Dose escalation study with 5 dose levels: DL1-1×10^7 cells/m2, DL2-3×10^7 cells/m2, and DL3-1×10^8 cells/m2, DL4- 2 to 3×10^8 cells/m2, DL5- 0.8 to 1×10^9 cells/m2
  Group A -HPVST cells Group B -lymphodepletion & nivolumab & HPVST cells.
  First, treatment in Group A will be completed for DL1 and DL2. Only if DL2 in Group A proves safe, Group B will be treated on DL2, DL3, DL4, and DL5.
  Group A will be treated at DL3, DL4, and DL5 only if there is excessive toxicity in cohorts treated with lymphodepletion.
  HPVSTs will be given by IV injection over 1-10 minutes through a peripheral or a central line on day 0.
  If patients have clinical benefit (as determined by symptoms, physical exam or radiological studies) & no significant toxicities, they may get up to 5 repeat infusions (for max total of 6 infusions) of HPVSTs at or below the same dose level.
  Other Names: HPVSTs
Drug: Cytoxan — 500mg/m^2/day x 3 days (on days -4, -3 and -2)
  Other Names: cyclophosphamide
  Arms: Group B
Drug: Fludarabine — 30mg/m^2/day x 3 days (on days -4, -3, and -2)
  Other Names: Fludara
  Arms: Group B
Biological: Nivolumab — 240mg every 2 weeks (+/- 3 days) starting on day -1
  Other Names: Opdivo
  Arms: Group B

SUMMARY:
Subjects have a type of cancer that has been associated with an infection with a virus called human papilloma virus (HPV). The cancer has come back, has not gone away after standard treatment or the subject cannot receive standard treatment.

This is a research study using special immune system cells called HPVST cells, a new experimental treatment.

Investigators want to find out if they can use this type of treatment in patients with HPV-cancers. They have discovered a way to grow large number of HPV-specific T cells from the blood of patients with HPV-cancers. They want to see if these special white blood cells, called HPVST cells, that will have been trained to kill HPV infected cells can survive in the blood and affect the tumor. They will also see if they can make the T cells more active against the HPV-cancers by engineering them to be resistant to the TGF-beta chemical that these HPV-cancers produce. They will grow these HPVST cells from the patient's blood.

The purpose of this study is to find the biggest dose of HPVSTs that is safe, to see how long they last in the body, to learn what the side effects are and to see if the HPVSTs will help people with HPV associated cancers.

If the treatment with HPVST cells alone proves safe (Group A), additional group of patients (Group B) will receive Nivolumab in addition to HPVST cells in a lymphodepleted environment. Nivolumab is an antibody therapy that helps T cells control the tumor and it is FDA approved for the treatment of certain types of cancers, including Hodgkin's lymphoma. Lymphodepletion will decrease the level of circulating T cells prior to infusion of HPVST cells, thereby giving them room to expand. The purpose of this part of the study is to find out if TGF-beta resistant HPVST cells in combination with Nivolumab are safe, how long they last in the body and if they are more effective than HPVST cells alone in controlling the tumor.

DETAILED DESCRIPTION:
HPV is found in the cancer cells of more than half the patients with certain types of cancer, suggesting that it may play a role in causing the cancer. The virus makes proteins in the tumor cells that should allow the diseased cells to be recognized and killed by a part of the body's own immune system called T cells. Unfortunately, tumors are able to avoid being killed by making molecules that turn off these T cells. So, the cancer cells infected by HPV are able to hide from the body's immune system and escape destruction.

The investigators have previously studied cancers caused by a different virus, called Epstein-Barr virus (EBV). These EBV-cancers are like HPV-cancers, since they turn off the T cells that would otherwise destroy them, and so can keep growing. They investigators have found, however, that if they removed the T cells from the blood of patients with EBV-cancers and grew them outside the body, they could increase the number and the activity of T cells directed against the tumors. When these T cells were given back to the patients, the T cells eliminated the cancers in over half the recipients. Investigators also found that they could engineer the T cells to be even more active against the EBV-cancer cells by making them resist an inhibitory chemical called TGF-beta, which is produced by these cancer cells.

Investigators will collect up to 390 mL of blood. Then they will use this blood to grow T cells. First they will grow them in a special type of cell called a dendritic cell, which stimulates the T cells. These dendritic cells will then be loaded with bits of proteins from the HPV virus called E6 and E7. These dendritic cells will be used to stimulate T cells. This stimulation trains the T cells to kill cells with the HPV proteins E6 and E7 on their surface. Next, the investigators will grow these HPV-specific T cells by more stimulation with dendritic cells and HPV proteins, and, when needed, a special type of cell called K562. These K562 cells were treated with radiation so they cannot grow.

To make these T cells resistant to the TGF-beta released by the tumor, investigators will put a new gene in them in the laboratory called a mutant TGF-beta receptor. In cells with this new gene, TGF-beta released by the tumor cells will not be able to bind to the mutant TGF-beta receptor on the T cell. Investigators hope this will improve the chances that after the T cells are injected they will be able to keep working and kill the tumor cells. This gene is added to the cells using a mouse retrovirus that has been changed to stop it from causing infections. Retroviruses enter the cell's DNA (genetic material) to make permanent changes to the cell. After making these cells, they will be frozen.

For treatment, the cells will be thawed and injected in a vein over 1 to 10 minutes. Initially, one dose of T cells will be given (which is considered day 0).

If, after the 1st infusion, there is a reduction in the size of the subject's cancer (or no increase) on CT or MRI scans as assessed by a radiologist, the subject can receive additional doses if it would be to his/her benefit, if s/he would like to receive more doses, and if there is enough product remaining to give any additional injections (at the same or a lower dose).

If treatment with HPVST cells alone proves safe, additional group of patients (Group B) will receive HPVST cells with nivolumab in lymphodepleted environment. One dose of the drug nivolumab is given one day before the HPVST cells are infused and then every 2 weeks for a total of four doses of nivolumab. Lymphodepletion will be given daily starting day -4 prior to administration of HPVSTs.

This is a dose escalation study. The dose the patient will get will depend on how many participants get the agent beforehand and how they react.

Investigators will follow the patient during and after the injections at predetermined time points which may require blood draws and other examinations.

ELIGIBILITY:
Inclusion Criteria:

PROCUREMENT

1. Diagnosis of a cancer for which the presence of a high risk HPV type has been documented in a biopsy sample
2. Cancer is:

   * recurrent or persistent after standard therapy
   * OR patient is unable to receive standard therapy
3. Karnofsky score ≥ 50%
4. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent

TREATMENT

1. Diagnosis of a cancer for which the presence of a high risk HPV type has been documented in a biopsy sample
2. Cancer is:

   * recurrent or persistent after standard therapy
   * OR patient is unable to receive standard therapy
3. Life expectancy ≥ 6 weeks.
4. Age ≥ 18 years.
5. Karnofsky score ≥ 50%
6. Bilirubin < 3 × upper limit of normal (ULN), AST < 5 × ULN, Hgb ≥ 7.0 g/dL
7. Pulse oximetry of > 90% on room air.
8. GFR > 30 mL/min calculated by the Cockcroft-Gault, MDRD study, or CKD-EPI creatinine equations, or equivalent.
9. ANC > 1.0/μL
10. Platelets > 75,000/μL
11. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent
12. Sexually active patients must be willing to utilize one of the more effective birth control methods during the study and for 6 months after the study is concluded. The male partner should use a condom.

Exclusion Criteria:

PROCUREMENT

1. Known HIV positivity.

TREATMENT

1. Currently receiving any investigational agents or have received any tumor vaccines or T cell antibodies within previous 4 weeks.
2. Severe intercurrent infection.
3. Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-09; Primary Completion 2026-01 (Estimated); Study Completion 2033-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicity (DLT) | 6 weeks
  DLT will be defined as any toxicity that is irreversible or life threatening, defined as the following, considered to be possibly, probably, or definitely related to the HPVST injection.
  1. Non-hematologic DLT is any grade 3 or grade 4 non-hematologic toxicity.
  2. Hematologic DLT is defined as any grade 4 hematologic toxicity.

SECONDARY OUTCOMES:
Overall response rate | 6 weeks
  To measure anti-tumor effects of HPV-specific T lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Ramos, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States